CLINICAL TRIAL: NCT01133977
Title: An Open-Label, Multicenter, Randomized, Phase Ib/II Study of E7080 (Lenvatinib) in Combination With Dacarbazine Versus Dacarbazine Alone as First Line Therapy in Patients With Stage IV Melanoma.
Brief Title: E7080 (Lenvatinib) in Combination With Dacarbazine Versus Dacarbazine Alone as First Line Therapy in Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-702
Record Dates: First submitted 2010-05-21; First posted 2010-05-31 (Estimated); Results first posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-08

CONDITIONS: Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — lenvatinib; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lenvatinib + Dacarbazine (Phase 1b) (Experimental): Participants received 16 mg, 20 mg or 22 mg lenvatinib once daily in combination with dacarbazine
  Interventions: Drug: Lenvatinib; Drug: Dacarbazine
- Lenvatinib + Dacarbazine (Phase 2) (Experimental): Participants received lenvatinib per the maximum tolerated dose (MTD) as determined in the Phase Ib of the study in combination with dacarbazine
  Interventions: Drug: Lenvatinib; Drug: Dacarbazine
- Dacarbazine (Phase 2) (Active Comparator): Participants received dacarbazine
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib tablets administered orally at doses of 16 mg, 20 mg, or 22 mg, once daily continuously over 3 weeks (21 days) during each 21-day cycle
  Other Names: E7080
  Arms: Lenvatinib + Dacarbazine (Phase 1b)
Drug: Lenvatinib — Lenvatinib 20 mg (MTD/recommended Phase 2 dose as determined in Phase 1b of the study) administered once daily continuously over 3 weeks (21 days) during each 21-day cycle
  Other Names: E7080
  Arms: Lenvatinib + Dacarbazine (Phase 2)
Drug: Dacarbazine — Dacarbazine (1000 mg/m2) infusion over 60 minutes on Day 1 of each 21-day cycle.
  Other Names: Dacarbazine (DTIC)-Dome

SUMMARY:
Primary:

* Phase Ib: To define the safety, tolerability and maximum tolerated dose (MTD) of lenvatinib administered in combination with dacarbazine.
* Phase II: To evaluate the safety and tolerability of lenvatinib administered in combination with dacarbazine, compared with dacarbazine alone.

Secondary:

-Phase II: To make a preliminary assessment of the efficacy of lenvatinib administered in combination with dacarbazine, compared with dacarbazine alone.

DETAILED DESCRIPTION:
Safety was assessed by monitoring and recording all treatment emergent adverse events (AEs) and serious adverse events (SAEs); regular monitoring of clinical laboratory parameters; periodic measurement of vital signs and electrocardiograms (ECGs); dose limiting toxicities; performance of physical examinations; concomitant medications and procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically-confirmed metastatic melanoma (Stage IV, American Joint Committee on Cancer (AJCC)).
2. No prior cytokine, chemotherapy, or targeted therapy for Stage IV melanoma.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
4. Life expectancy greater than or equal to 3 months.
5. At least 1 site of measurable disease by RECIST 1.1.
6. Adequate hematologic, renal, liver, and coagulation system function as defined by laboratory values performed within 21 days prior to initiation of dosing.
7. Blood pressure must be well-controlled (less than or equal to 140/90 mmHg at screening) with or without antihypertensive medication. Patients must have no history of hypertensive crisis or hypertensive encephalopathy.

Exclusion Criteria:

1. Known central nervous system (CNS) lesions, except for asymptomatic, nonprogressive, treated brain metastases. Treatment for brain metastases must have been completed at least 4 weeks prior to Day 1 and may include whole brain radiotherapy (WBRT), radiosurgery [RS; Gamma Knife, linear accelerator (LINAC), or equivalent] or a combination as deemed appropriate by the treating physician. Dexamethasone must be discontinued at least 3 weeks prior to Day 1. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
2. Lactate dehydrogenase greater than or equal to 2.0 x upper limit of normal (ULN).
3. Subjects with proteinuria greater than 1+ on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria. Subjects with 24-hour urine protein greater than or equal to 1 g/24 hours will be ineligible.
4. Pregnant, breast-feeding, or refusing double barrier contraception, oral contraceptives or avoidance of pregnancy measures.
5. Other active malignancy.
6. History of or known carcinomatous meningitis.
7. History of or known ocular melanoma.
8. Are currently receiving any other treatment for the tumor (including palliative radiotherapy) aside from control of symptoms.
9. Received treatment in another clinical study within the 30 days prior to commencing study treatment or patients who have not recovered from side effects of an investigational drug to grade less than or equal to 1, except for alopecia.
10. Received radiotherapy within the 30 days prior to commencing study treatment or have not recovered from side effects of all radiation-related toxicities to grade less than or equal to 1, except for alopecia.
11. Serious non-healing wound, ulcer, bone fracture, or have undergone a major surgical procedure, open biopsy, or significant traumatic injury within the 28 days prior to commencing study treatment. Minor surgery such as Portacath placement or skin biopsy is permitted if greater than or equal to 7 days have passed.
12. History of bleeding diathesis or coagulopathy.
13. Current use of anti-coagulants such as Vitamin K antagonists, unfractionated heparin, or low molecular weight heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2010-04; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Harish, Study Director — Quintiles, Inc.
Locations (23):
- United States (5):
  - Hagerstown, Maryland
  - Albany, New York
  - Greenville, South Carolina
  - Dallas, Texas
  - Norfolk, Virginia
- Germany (3):
  - Berlin
  - Heidelberg
  - München
- Italy (5):
  - Bari
  - Milan
  - Milian
  - Napoli
  - Siena
- Spain (3):
  - Barcelona
  - Madrid
  - Valenica
- United Kingdom (7):
  - Dorset
  - Glasgow
  - Manchester
  - Metropolitan Borough of Wirral
  - Middlesex
  - Oxford
  - Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 16 participants were enrolled in the Phase 1b portion of the study; all 16 participants received study treatment. A total of 82 participants were randomized in the Phase 2 portion of the study and a total of 81 participants received treatment. In the Darcarbazine arm, one participant withdrew consent prior to receiving study treatment.
Groups:
- 16 mg Lenvatinib + Dacarbazine (Phase 1b): Participants received 16 mg lenvatinib once daily continuously over 3 weeks (21 days) during each cycle in combination with dacarbazine (1000 mg/m2) on Day 1 of each 21-day cycle upto eight 21-day cycles (24 weeks) or more if participants experience clinical benefit
- 20 mg Lenvatinib + Dacarbazine (Phase 1b); 20 mg Lenvatinib + Dacarbazine (Phase 2): Participants received 20 mg lenvatinib once daily continuously over 3 weeks (21 days) during each cycle in combination with dacarbazine (1000 mg/m2) on Day 1 of each 21-day cycle upto eight 21-day cycles (24 weeks) or more if participants experience clinical benefit
- 22 mg Lenvatinib + Dacarbazine (Phase 1b): Participants received 22 mg lenvatinib once daily continuously over 3 weeks (21 days) during each cycle in combination with dacarbazine (1000 mg/m2) on Day 1 of each 21-day cycle upto eight 21-day cycles (24 weeks) or more if participants experience clinical benefit
- Dacarbazine (Phase 2): Participants received dacarbazine (1000 mg/m2) on Day 1 of each 21-day cycle upto eight 21-day cycles (24 weeks) or more if participants experience clinical benefit
Period: Overall Study
Arm/Group | 16 mg Lenvatinib + Dacarbazine (Phase 1b) | 20 mg Lenvatinib + Dacarbazine (Phase 1b) | 22 mg Lenvatinib + Dacarbazine (Phase 1b) | 20 mg Lenvatinib + Dacarbazine (Phase 2) | Dacarbazine (Phase 2)
Started | 3 (Treated) | 7 (Treated) | 6 (Treated) | 42 (Treated) | 39 (Treated)
Completed | 0 | 0 | 0 | 3 | 1
Not Completed | 3 | 7 | 6 | 39 | 38
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Death | 1 | 1 | 1 | 7 | 3
Not completed — Started a New Line of Therapy | 2 | 6 | 4 | 25 | 33
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 1

BASELINE CHARACTERISTICS:
Population: A total of 40 participants were randomized in Dacarbazine (Phase 2) arm but only 39 participants received study drug and were included in the safety analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | 16 mg Lenvatinib + Dacarbazine (Phase 1b) | 20 mg Lenvatinib + Dacarbazine (Phase 1b) | 22 mg Lenvatinib + Dacarbazine (Phase 1b) | 20 mg Lenvatinib + Dacarbazine (Phase 2) | Dacarbazine (Phase 2) | Total
Number analyzed (Participants) | 3 | 7 | 6 | 42 | 39 | 97
Age, Customized [Number; unit: Participants]
  18 years and older | 3 | 7 | 6 | 42 | 39 | 97
Sex/Gender, Customized [Number; unit: participants]
  Male | 3 | 2 | 4 | 25 | 23 | 57
  Female | 0 | 5 | 2 | 17 | 16 | 40

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) of Lenvatinib Administered in Combination With Dacarbazine (for Phase 1b)
Description: DLTs were defined as clinically significant adverse events (AEs) occurring less than or equal to 21 days after commencing study treatment and considered by the Investigator to be possibly or probably related to study treatment.
Time Frame: From Day 1 through 21 days (one cycle)
Population: Safety Analysis Set: All participants enrolled in the Phase 1b portion of this study, except for those who (i) dropped out of the study prior to receiving any study drug, or (ii) were without any safety assessment following the first dose of study drug.
Measure: Number; unit: Participants with DLT
Arm/Group | 16 mg Lenvatinib + Dacarbazine (Phase 1b) | 20 mg Lenvatinib + Dacarbazine (Phase 1b) | 22 mg Lenvatinib + Dacarbazine (Phase 1b)
Number analyzed (Participants) | 3 | 7 | 6
Participants with DLT
  Participants with DLTs | 0 | 1 | 2
  Grade 3 hypertension | 0 | 1 | 1
  Grade 3 febrile neutropenia | 0 | 0 | 1
  Grade 3 thrombocytopenia | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Adverse Events/Serious Adverse Events (AEs/SAEs)
Description: Safety assessments consisted of monitoring and recording all AEs, including all Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v. 4.0) grades, and SAEs; regular monitoring of hematology, blood chemistry, and urine values; periodic measurement of vital signs and electrocardiograms (ECGs); and performance of physical examinations. Details of AEs and SAEs are provided in the reported adverse event section.
Time Frame: From signing of informed consent up to 30 days after the last dose, up to approximately 2 years
Population: Safety Analysis Set: All participants enrolled in the Phase 1b and Phase 2 portion of this study, except for those who (i) dropped out of the study prior to receiving any study drug, or (ii) were without any safety assessment following the first dose of study drug.
Measure: Number; unit: Participants
Arm/Group | 16 mg Lenvatinib + Dacarbazine (Phase 1b) | 20 mg Lenvatinib + Dacarbazine (Phase 1b) | 22 mg Lenvatinib + Dacarbazine (Phase 1b) | 20 mg Lenvatinib + Dacarbazine (Phase 2) | Dacarbazine (Phase 2)
Number analyzed (Participants) | 3 | 7 | 6 | 42 | 39
Participants
  AEs | 3 | 7 | 6 | 40 | 31
  SAEs | 2 | 4 | 2 | 16 | 1

3. Secondary Outcome: Progression Free Survival (PFS) (for Phase 2)
Description: PFS was defined as the time from the date of randomization of a participant until (1) the date of first documented progression of such participant's disease based on Investigator assessments according to Response Evaluation Criteria In Solid Tumors (RECIST v. 1.1) or (2) the date of such participant's death due to any cause. Progression was defined as at least a 20% increase or 5 mm increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions, based on Investigator assessment according to RECIST 1.1. If missing assessments, imputed dates were used in the analysis.
Time Frame: From the date of randomization until the date of disease progression or death (whichever was earlier) or up to approximately 2 years
Population: All randomized participants who received at least one dose of study drug without major protocol eligibility violations were included in the Modified Intent-to-Treat (MITT) Analysis Set.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | 20 mg Lenvatinib + Dacarbazine (Phase 2) | Dacarbazine (Phase 2)
Number analyzed (Participants) | 40 | 37
Weeks | 19.1 [9.57 to 25.57] | 7.0 [5.57 to 15.57]
Statistical Analysis 1: Comparison: 20 mg Lenvatinib + Dacarbazine (Phase 2) vs Dacarbazine (Phase 2); The current study was not powered or designed to determine superiority of the '20 mg Lenvatinib + Dacarbazine (Phase 2)' arm compared with 'Dacarbazine (Phase 2) ' arm; Test type: Superiority or Other; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.23 to 0.75]

4. Other Pre Specified Outcome: Time to Progression (TTP) (for Phase 2)
Description: TTP, defined as the time from the date of randomization until the date of progressive disease.
Time Frame: From the date of randomization until disease progression or death or up to approximately 2 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Overall Survival (OS) (for Phase 2)
Description: OS, defined as the time from the date of randomization until the date of death. Few events of deaths (9 events in the Lenvatinib + Dacarbazine arm and 4 events in the Dacarbazine arm) were reported to calculate the median OS or to draw conclusions regarding the OS.
Time Frame: From the date of randomization until death or up to approximately 2 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Overall Response Rate (ORR) (for Phase 2)
Description: ORR, defined as percentage of participants with best confirmed response (complete response [CR] or partial response [PR]). A confirmatory scan was required after no less than 4 weeks and no later than 8 weeks, starting on the date that the response was first recorded.
Time Frame: From the date of randomization until disease progression or death or up to approximately 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to 30 days after the last dose, up to approximately 2 years.
Description: Treatment emergent adverse events (TEAEs), defined as an AE that started/increased in severity on/after the first dose of study drug up to 30 days after final dose of study drug are reported.
Arm/Group | 16 mg Lenvatinib + Dacarbazine (Phase 1b) | 20 mg Lenvatinib + Dacarbazine (Phase 1b) | 22 mg Lenvatinib + Dacarbazine (Phase 1b) | 20 mg Lenvatinib + Dacarbazine (Phase 2) | Dacarbazine (Phase 2)
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/7 | 2/6 | 16/42 | 1/39
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 6/6 | 40/42 | 31/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 16 mg Lenvatinib + Dacarbazine (Phase 1b) (N=3) | 20 mg Lenvatinib + Dacarbazine (Phase 1b) (N=7) | 22 mg Lenvatinib + Dacarbazine (Phase 1b) (N=6) | 20 mg Lenvatinib + Dacarbazine (Phase 2) (N=42) | Dacarbazine (Phase 2) (N=39)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
White Blood Cell Count Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Intertrigo Candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Partial Seizures (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Breast Swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Physical Disability (Social circumstances) | 0 | 0 | 0 | 1 | 0
Hypertention (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 16 mg Lenvatinib + Dacarbazine (Phase 1b) (N=3) | 20 mg Lenvatinib + Dacarbazine (Phase 1b) (N=7) | 22 mg Lenvatinib + Dacarbazine (Phase 1b) (N=6) | 20 mg Lenvatinib + Dacarbazine (Phase 2) (N=42) | Dacarbazine (Phase 2) (N=39)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 4 | 4
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2 | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 3 | 2 | 10 | 4
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 3 | 2 | 5 | 1
CONDUCTION DISORDER (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 2 | 0 | 7 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 3 | 1 | 6 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 4 | 1 | 14 | 14
DIARRHOEA (Gastrointestinal disorders) | 1 | 4 | 2 | 13 | 6
DIVERTICULUM (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 1 | 0 | 5 | 1
DYSPEPSIA (Gastrointestinal disorders) | 1 | 2 | 0 | 8 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 5 | 4 | 16 | 11
ORAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 3 | 1 | 2 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
VOMITING (Gastrointestinal disorders) | 2 | 4 | 0 | 10 | 4
ASTHENIA (General disorders) | 1 | 3 | 1 | 7 | 7
CATHETER SITE PAIN (General disorders) | 0 | 1 | 0 | 1 | 0
CHILLS (General disorders) | 0 | 1 | 0 | 0 | 3
FATIGUE (General disorders) | 2 | 5 | 2 | 10 | 7
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1 | 0 | 0 | 0
INFUSION SITE REACTION (General disorders) | 0 | 0 | 1 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 0 | 0 | 0 | 3 | 0
PAIN (General disorders) | 0 | 2 | 1 | 4 | 0
PYREXIA (General disorders) | 0 | 2 | 0 | 7 | 1
CONJUNCTIVITIS VIRAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CYSTITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0
FOLLICULITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1 | 0 | 1 | 0
HORDEOLUM (Infections and infestations) | 0 | 1 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 0 | 2
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 3 | 4
ORAL FUNGAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
RHINITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 2
SINUSITIS (Infections and infestations) | 0 | 1 | 0 | 2 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0 | 4 | 3
BAROTRAUMA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 3 | 0 | 5 | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 2 | 0 | 3 | 2
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 2
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1 | 1 | 1 | 0
BLOOD URIC ACID INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 3 | 2
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 2 | 0 | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 0 | 2 | 0 | 3 | 1
WEIGHT DECREASED (Investigations) | 2 | 1 | 0 | 3 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 5 | 0 | 10 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 7 | 3
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 5 | 2
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
SUPERFICIAL SPREADING MELANOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 1 | 0 | 2 | 1
DYSAESTHESIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 1 | 1 | 0 | 1 | 3
HEADACHE (Nervous system disorders) | 1 | 4 | 1 | 4 | 3
LETHARGY (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
MIGRAINE (Nervous system disorders) | 0 | 0 | 0 | 3 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
ANXIETY (Psychiatric disorders) | 0 | 1 | 0 | 3 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0
DISORIENTATION (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 1 | 1 | 1 | 1
DYSURIA (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 1 | 0 | 8 | 2
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
BREAST DISORDER (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
MENSTRUATION IRREGULAR (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 5 | 4
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 11 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1 | 1
PHARYNGEAL ERYTHEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
ACNE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3 | 2
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 4 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 3 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
FLUSHING (Vascular disorders) | 0 | 1 | 0 | 1 | 2
HYPERTENSION (Vascular disorders) | 1 | 6 | 5 | 20 | 2
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 0 | 1 | 0 | 0
HYPOTENSION (Vascular disorders) | 0 | 0 | 1 | 4 | 0
PHLEBITIS (Vascular disorders) | 0 | 1 | 0 | 0 | 0
VASCULITIS (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other